CLINICAL TRIAL: NCT05047185
Title: A Phase II, Double-blind, Placebo-controlled, Randomized, Dose-ranging, Parallel Group Study to Evaluate the Safety and Efficacy of PHA-022121 Administered Orally for Prophylaxis Against Angioedema Attacks in Patients With Hereditary Angioedema Due to C1-Inhibitor Deficiency (Type I or Type II)
Brief Title: Dose-ranging Study of Oral PHA-022121 for Prophylaxis Against Angioedema Attacks in Patients With Hereditary Angioedema Type I or Type II
Acronym: HAE CHAPTER-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pharvaris Netherlands B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PHA022121-C301; 2021-000227-13 (EudraCT Number)
Record Dates: First submitted 2021-09-07; First posted 2021-09-17 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Hereditary Angioedema; Hereditary Angioedema Type I; Hereditary Angioedema Type II; Hereditary Angioedema Types I and II; Hereditary Angioedema Attack; Hereditary Angioedema With C1 Esterase Inhibitor Deficiency; Hereditary Angioedema - Type 1; Hereditary Angioedema - Type 2; C1 Esterase Inhibitor Deficiency; C1 Inhibitor Deficiency
Keywords: HAE; HAE Type I; HAE Type II; Oral Treatment; Bradykinin B2 Receptor Antagonist; PHVS416; PHA121; Prophylaxis; Deucrictibant
MeSH Terms: conditions — Angioedemas, Hereditary; Hereditary Angioedema Types I and II

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1: Low dose (Experimental): BID low dose of deucrictibant
  Interventions: Drug: Deucrictibant low dose
- Part 1: High dose (Experimental): BID high dose of deucrictibant
  Interventions: Drug: Deucrictibant high dose
- Part 1: Placebo (Placebo Comparator): BID placebo
  Interventions: Drug: Placebo
- Part 2: Open-label (Experimental): BID high dose of deucrictibant
  Interventions: Drug: Deucrictibant high dose

INTERVENTIONS:
Drug: Deucrictibant low dose — Deucrictibant softgel capsules for oral use (PHVS416)
  Arms: Part 1: Low dose
Drug: Deucrictibant high dose — Deucrictibant softgel capsules for oral use (PHVS416)
  Arms: Part 1: High dose; Part 2: Open-label
Drug: Placebo — Matching placebo capsules for oral use
  Arms: Part 1: Placebo

SUMMARY:
This study evaluates the safety and efficacy of PHA-022121 administered orally for prophylaxis against angioedema attacks in patients with hereditary angioedema (HAE). The study consists of 2 parts, with patients completing participation in Part 1 prior to initiation of treatment in Part 2. Part 1 of the study has 3 parallel arms and approximately 30 patients will be equally randomized to one of two dose regimens of PHA-022121 or matching placebo. Patients will continue to the single open-label arm in Part 2 of the study after completion of Part 1. The screening period is up to 8 weeks and the treatment periods are 12 weeks (Part 1) and 30 months (Part 2) in duration.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent form
* Diagnosis of HAE type I or II
* Documented history of at least 3 HAE attacks within the last 3 consecutive months prior to screening, or a minimum of 2 HAE attacks during the screening period
* Reliable access and experience to use standard of care acute attack medications

Exclusion Criteria:

* Pregnancy or breast-feeding
* Clinically significant abnormal electrocardiogram
* Any other systemic disease or significant disease or disorder that would interfere with the patient's safety or ability to participate in the study
* Use of C1-esterase inhibitor, oral kallikrein inhibitors, attenuated androgens, anti-fibrinolytics, or monoclonal HAE therapy within a defined period prior to enrolment
* Abnormal hepatic function
* Abnormal renal function
* History of alcohol or drug abuse within defined period, or current evidence of substance dependence or abuse
* Participation in any other investigational drug study within defined period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Number of investigator-confirmed HAE attacks | Day 0 to Day 84

SECONDARY OUTCOMES:
Number of investigator-confirmed moderate or severe HAE attacks during the treatment period | Day 0 to Day 84
Number of investigator-confirmed HAE attacks requiring acute treatment during the treatment period | Day 0 to Day 84
Number of patients achieving reduction in attack rate during the treatment period relative to baseline | Day 0 to Day 84
Number of patients that are attack-free during the treatment period | Day 0 to Day 84
Number and proportion of days with angioedema symptoms during the treatment period | Day 0 to Day 84
Time to first investigator-confirmed HAE attack in the treatment period | Day 0 to Day 84
Number of investigator-confirmed HAE attacks resulting in a visit to the emergency department or an admission to hospital | Day 0 to Day 84
Number of investigator-confirmed angioedema attacks during the treatment period in Part 2. | Day 84 to Day 938
Number of investigator-confirmed moderate or severe angioedema attacks during the treatment period in Part 2. | Day 84 to Day 938
Number of investigator-confirmed angioedema attacks requiring acute treatment during the treatment period in Part 2. | Day 84 to Day 938
Incidence of HAE attacks during the treatment period in Part 2 (attack rate trend over time). | Day 84 to Day 938
Number and proportion of days with angioedema symptoms during the treatment period in Part 2. | Day 84 to Day 938

CONTACTS AND LOCATIONS:
Overall Officials: Marc Riedl, MD, Principal Investigator — UC San Diego, La Jolla, California, United States; Emel Aygören-Pürsün, MD, Principal Investigator — University Hospital Frankfurt - Goethe University, Frankfurt, Germany
Locations (19):
- United States (3):
  - Study site, Birmingham, Alabama
  - Study site, Paradise Valley, Arizona
  - Study site, St Louis, Missouri
- Study Site, Vienna, Austria
- Study site, Sofia, Bulgaria
- Canada (2):
  - Study site, Ottawa, Ontario
  - Study site, Montreal, Quebec
- Germany (2):
  - Study site, Berlin
  - Study site, Frankfurt
- Study site, Dublin, Ireland
- Italy (3):
  - Study site, Padua, PD
  - Study site, Milan
  - Study site, Palermo
- Study site, Krakow, Poland
- United Kingdom (5):
  - Study site, Brighton, England
  - Study site, Bristol, England
  - Study site, Cambridge, England
  - Study site, London, England
  - Study site, Southampton, England

IPD SHARING:
Plan to Share IPD: No